CLINICAL TRIAL: NCT06872255
Title: A Prospective Pilot Trial of Per-oral Endoscopic Myotomy (POEM) in Patients with Postfundplication Dysphagia (VADYSMA Trial)
Brief Title: Per-oral Endoscopic Myotomy (POEM) in Patients with Postfundplication Dysphagia
Acronym: VADYSMA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Collaborators: University Hospital Trnava (Network); St. Anne's University Hospital Brno, Czech Republic (Other)
Responsible Party: Principal Investigator, Prof. Jan Martinek, MD, PhD, AGAF, Head of Gastroenterology and hepatology department, St. Anne's University Hospital Brno, Czech Republic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VADYSMA
Record Dates: First submitted 2025-02-10; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Dysphagia; Dysphagia, Esophageal; Healthy
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Patients with refractory (> 6 months) and severe dysphagia after fundoplication procedure defined as an Eckardt score ≥3 and Mellow - Pinkas score ≥2 at baseline, with proven obstruction of gastroesofageal junction (EGJOO)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- POEM arm (Experimental): Patients, who will undergo peroral endoscopic myotomy for postfundoplication dysphagia
  Interventions: Procedure: Per Oral Endoscopic Myotomy (POEM)

INTERVENTIONS:
Procedure: Per Oral Endoscopic Myotomy (POEM) — All procedures will be performed by an experienced endoscopist, with a sufficient experience in "third space" endoscopy (at least 100 POEMs) under general anesthesia (internal preoperative examination is necessary) with a high-definition endoscope, fitted with a plastic distal attachment. Before the procedure, the patients will be administered intravenous antibiotics. Exclusively CO2 will be used for insufflation. POEM will be performed in a similar way as in patients with achalasia - the procedure consists of 4 steps: (1) mucosal incision and tunnel entry, (2) submucosal tunneling, (3) myotomy, and (4) closure of the mucosal entry with endoscopic clips or other closure devices. Perioperative protocol might differ according the usual way of performing POEM in a given center.

SUMMARY:
Laparoscopic fundoplication represents the standard antireflux procedure, when conservative measures fail. However, any type of fundoplication may be accompanied by adverse events. Postfundoplication dysphagia (PFD) may hamper results of anti-reflux surgery. Endoscopic pneumatic dilation has been considered as the first line treatment option for persistent PFD. However, studies have not confirmed its effectiveness in this indication. Peroral endoscopic myotomy (POEM) became a standard treatment for the management of esophageal achalasia and moreover has also been assessed in a small cohort of patients with refractory PFD and some patients achieved significant treatment success. We plan to perform a prospective international cohort multicenter study assessing the efficacy of POEM in patients with persistent and severe PFD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients after laparoscopic fundoplication procedure by Nissen (total, 360°), Dor (anterior, 180°) or Toupet (posterior, 270°) for gastroesophageal reflux disease no later than 10 years before enrolment.
2. Refractory (> 6 months) and severe dysphagia after fundoplication procedure defined as an Eckardt score ≥3 and Mellow - Pinkas score ≥2 at baseline.
3. X-ray (contrasted radiographic examination of the esophagus) characterized by both: a.) tapered narrowing of the distal esophagus and GEJ; b.) partial/total stagnation of the contrast solution above the GEJ
4. Endoluminal planimetry: EGJ-DI < 3 mm2/mmHg (with 40ml)
5. Age above 18 years
6. Signed informed consent form

Exclusion Criteria:

1. No previous attempt with at least one prokinetic drug
2. Previous esophageal myotomy (open, laparoscopic or endoscopic)
3. Primary esophageal motility disorder (achalasia etc.)
4. Active erosive esophagitis
5. Active peptic ulcer disease
6. Esophageal stricture (peptic, malignant, other)
7. Partial or complete supradiaphragmatic migration of the wrap and/or stomach (Hinder Type III - IV), Large hiatal hernia more than 5 cm
8. Known eosinophilic esophagitis
9. Severe coagulopathy
10. Esophageal or gastric varices
11. Advanced liver cirrhosis (Child B or Child C)
12. Pregnancy or puerperium
13. Malignant or pre-malignant esophageal diseases (dysplasia): patients with a history of such disease after its cure are eligible for enrolment
14. Any other condition, which in the opinion of the investigator would interfere with study requirements
15. Known gastroparesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy and safety of POEM in patients with postfundoplication dysfagia | 6 months
  The primary outcome will be proportion of patients with treatment success defined as Eckardt score ≤ 2 and its decrease by at least 1 point after POEM at 6 months

SECONDARY OUTCOMES:
Eckardt score | At baseline and after 3, 6 and 12 months
  The Eckardt score is the grading system used for the evaluation of severity of symptoms in patients with esophageal achalasia. Four symptoms are assessed (dysphagia, regurgitation, chest pain and weight loss) and their severity ranges from 0 (no symptom) to 3 (with every meal). Total score is their sum and ranges from 0 to 12
Mellow - Pinkas score | At baseline and after 3, 6 and 12 months
  The Mellow - Pinkas score is used to assess dysphagia grade before and after the interventions. Total score ranges from 0 to 3 (0 = able to eat normal diet, 1 = able to swallow some solid foods, 2 = able to swallow only semi solid foods, 3 = able to swallow liquids only)
PAGI-QOL score (Patient Assessment of Upper Gastrointestinal Disorders-Quality of Life) | At baseline and after 3, 6 and 12 months
  The PAGI-QoL questionnaire contains of 30 items with five subscales: (1) daily activities; (2) clothing; (3) diet/food habits; (4) relationship; and (5) psychological well-being and distress. Each item is scored on a 6-point Likert scale, with response options ranging from 0 (none) to 5 (severe problem all of the time). Subscale scores are calculated by averaging the item responses. A total score is calculated by averaging subscale scores. Higher score means impairment in quality of life.
GERD-RHQL score (Gastroesophageal Reflux Disease Health-related Quality of Life) | At baseline and after 3, 6 and 12 months
  The GERD-HRQL questionnaire was developed and validated to measure changes of typical GERD symptoms such as heartburn and regurgitation in response to surgical or medical treatment. Higher (greater) possible score means worst symptoms - ranging from 0 to 75.
Integrated Relaxation Pressure (IRP) | At baseline and after 6 months
  High resolution manometry - Median IRP recorded from 10 supine swallows, measured in mmHg. A value >15 mmHg indicates EGJ outflow obstruction.
Endoluminal planimetry (Endoflip) | At baseline and after 6 months
  Pyloric distensibility measured by impedance planimetry (EndoFLIP device)
Esophagogram | At baseline and after 6 months
  Esophagogram provides valuable information of the fundoplication, better appreciate a paraesophageal hernia and information on esophageal emptying.
  Patients will be advised overnight fasting prior to timed barium esophagogram. A contrast agent (e.g. barium, usually 100 to 250 mL) is ingested orally within 15-20 seconds. Left posterior oblique X-ray will be taken 2 and 5 minutes after contrast agent ingestion. Maximum esophageal width and column hights will be recorded at 2 and 5 minutes.
Eckardt score | At and after 3 and 12 months
  The Eckardt score is used to assess the severity of achalasia symptoms. It is based on the four main symptoms of achalasia: dysphagia, regurgitation, chest pain and weight loss. Each symptom has four levels of severity: none = 0 point, occasional = 1 point, daily = 2 points, each meal = 3 points. The sum of the points gives the final score. Final score scale: 0 (best) - 12 (worst). Treatment success is defined as a decrease of Eckardt score by at least 1 point and an overall Eckardt score ≤ 2.
GERD | At baseline and after 3, 6 and 12 months
  Presence of reflux esophagitis based on endoscopy findings.
Esophageal 24h-Hour pH metry | At 3 months after procedure
  An esophageal pH test measures how often stomach acid enters to the esophagus. It also measures how long the acid stays there. The test involves placing a catheter into the esophagus. The catheter or device will measure an acid level (known as pH level) for 24 hours. Post-POEM Esophageal acid exposure (DeMeester score, proportion of time with pH below 4)After
PPI/H2 antagonists | At baseline and after 3, 6 and 12 months
  PPI's and/or H2 antagonists use before and after procedure (POEM).

CONTACTS AND LOCATIONS:
Locations (2):
- St. Anne's University Hospital Brno, Czech Republic, Brno, Czechia
- University Hospital Trnava, Trnava, Slovakia